CLINICAL TRIAL: NCT01945203
Title: The Relationship Between Aortic Pulse Wave, Aortic Calcification and Peripheral Artery Occlusion Disease in Peritoneal Dialysis Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201105097RC
Record Dates: First submitted 2013-09-09; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: End-stage Renal Disease; Peritoneal Dialysis; Aortic Calcification; Peripheral Artery Occlusion; Cardiovascular Disease
Keywords: Calcification; aortic pulse wave velocity; peripheral artery occlusion disease; peritoneal dialysis; metabolic syndrome
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases; Calcinosis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, 8ml/patient
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PD-ABI: 1. Patients at National Taiwan University Hospital (NTUH)
  2. Patients who have received PD more than 3 months
  3. Patients who sign the informed consents
  4. Patients who aged between 20-90 years.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of mortality in patients with end-stage renal disease (ESRD), which means that it is important to find out risk factors of CVD in order to prevent or treat it. In recent years, there has been more and more recognition of a very high prevalence of CV calcification in the ESRD population. Many observational cohort studies have shown that CV calcification in these patients can predict mortality, CV mortality and morbidity. Electrolyte imbalance is easily found in the ESRD patients which may result in vessel calcification. Calcification leads to arterial stenosis and increasing arterial stiffness and then heart afterload, both contribute to the development of CVD. Besides, metabolic syndrome, insulin resistance, and dyslipidemia pave the way for a chronic, immune-mediated vascular inflammation and cardiovascular disease. These factors are prevalent in ESRD patients, which would also cause arterial stiffness. Arterial stiffness and stenosis would increase the risk of CV events and mortality. Aortic pulse wave velocity is strongly associated with the presence and extent of atherosclerosis and constitutes a forceful marker and predictor of cardiovascular risk. At the same time, high prevalence of peripheral artery occlusion disease (PAOD) should also be found while arterial stiffness and stenosis, which would increase the condition of infection and gangrene. Thus, life safety and quality would be influenced severely and early detection might prevent future amputation. As compared with HD or pre-dialysis patients, uremic patients treated with PD have a higher risk for metabolic syndrome. Therefore, more studies to evaluate the condition of arterial stiffness and PAOD, especially in PD patients, are needed for future management and preventions of CV related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at National Taiwan University Hospital (NTUH)
2. Patients who have received PD more than 3 months
3. Patients who sign the informed consents

Exclusion Criteria:

1. Patients who refuse to sign informed consents
2. Patients who refuse to draw additional blood for research

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the associations between aortic pulse wave, ankle-brachial index, aortic calcification and blood/serum biochemical markers, such as MPO, MMP-9, IL-6, adiponectin, TNF-alpha, of the patients in prevalent peritoneal dialysis patients. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital (NTUH), Taipei, Taiwan, Taiwan